CLINICAL TRIAL: NCT03932149
Title: The Effect of Intermittent Theta Burst Stimulation (iTBS) in Patients With Alcohol Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JDu-007
Record Dates: First submitted 2019-04-17; First posted 2019-04-30 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-04

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Intermittent Theta Burst Stimulation; Alcohol Dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Real stimulation
  Interventions: Device: Intermittent Theta Burst Stimulation (iTBS)
- Control Group (Sham Comparator): Sham stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation (iTBS) — The target is left DLPFC and the iTBS protocol is: 70% of RMT; triplet 50 Hz bursts, repeated at 5 Hz; 2s on and 8s off; 600 pulses a session.
  Arms: Experimental Group
Device: Sham stimulation — The target is right DLPFC and the sham stimulation protocol is: triplet 50 Hz bursts, repeated at 5 Hz; 2s on and 8s off; 600 pulses a session.
  Arms: Control Group

SUMMARY:
The aim of this trial is to investigate the efficacy of left DLPFC iTBS in a population of alcohol use disorder patients, compared with the sham iTBS. Moreover, this trial will conduct follow-up assessments to evaluate whether its efficacy can sustain for a long time if it is effective.

DETAILED DESCRIPTION:
Alcohol abuse and alcohol use disorder are important major health issues in our modern society. However, the treatment of alcohol addiction is currently limited to the treatment of acute withdrawal symptoms, but lacks effective interventions to reduce craving and prevent relapse. In an attempt to improve the treatment of substance dependence, non-invasive neuromodulation has gained attention as a new potential treatment option. The aim of this trial is to investigate the efficacy of left DLPFC iTBS in a population of alcohol use disorder patients, compared with the sham iTBS. Moreover, this trial will conduct follow-up assessments to evaluate whether its efficacy can sustain for a long time if it is effective.

ELIGIBILITY:
Inclusion Criteria:

* a DSM-5 diagnosis of alcohol use disorder
* age between 18 and 65
* can return to the research center for successive visits.

Exclusion Criteria:

* severe cognitive impairment
* current DSM-5 diagnosis of schizophrenia or another psychotic disorder
* current other substance abuse (except nicotine)
* severe organic diseases
* rTMS contraindications (such as a history of epileptic seizures, metal implants near the head).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Craving change | baseline, after the intervention, and 3 months after the intervention
  Craving will be measured by visual analogue scale(VAS), participants specify their level of craving by indicating a position along a continuous line between two end-points, score ranges from 0 to 10, 0 refers to the lowest level of craving, 10 refers to the highest level of craving.

SECONDARY OUTCOMES:
The abstinence rate after the treatment | after the intervention, and 3 months after the intervention
  The abstinence rate defined as the number of abstinent days in the three months after the last simulation session
Change of depression | bbaseline, after the 2-weeks intervention, and 6 months after the intervention
  The decrease of Beck Depression Inventory (BDI) scores, a 21-question multiple-choice self-report inventory to measure the severity of depression .
Change of anxiety | baseline, after the 2-weeks intervention, and 6 months after the intervention
  The decrease of Beck Anxiety Inventory (BAI) scores, a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety.
Change of impulsiveness | baseline, after the 2-weeks intervention, and 6 months after the intervention
  The decrease of Barratt impulsiveness scale (BIS) scores，including 30 items.
Change of impulse control | baseline, after the 2-weeks intervention, and 6 months after the intervention
  The decrease of stop signal reaction time （SSRT） in the stop signal task.
Change of cognitive function | baseline, after the 2-weeks intervention, and 6 months after the intervention
  The increase of Cogstate scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yuan C, Su H, Chen T, Voon V, Du J. The Effect of Intermittent Theta Burst Stimulation (iTBS) in Patients With Alcohol Use Disorder: Study Protocol for a Randomized Controlled Trial. Front Psychiatry. 2020 Mar 10;11:210. doi: 10.3389/fpsyt.2020.00210. eCollection 2020. PMID 32218749